CLINICAL TRIAL: NCT04807998
Title: Risk Factors for Pediatric Emergence Agitation and Post-operative Pain Following Maxillofacial Surgery and Analysis of Serum or Urine Metabonomics in Children With Agitation-An Exploratory Study
Brief Title: Risk Factors for Pediatric Emergence Agitation and Analysis of Serum or Urine Metabonomics in Children With Agitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, vice-director, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: SH9H-2020-T149
Record Dates: First submitted 2021-02-21; First posted 2021-03-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Emergence Agitation; Pain; Metabolomics
Keywords: pediatric emergence agitation; postoperative Pain; metabolomics
MeSH Terms: conditions — Emergence Delirium; Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients' blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group EA: Serum and Urine samples were collected before anesthesia and immediately after surgery from children who enrolled in part I and undergoing the adenoidectomy or adenotonsillectomy. A PAED score of 12 or greater was defined as EA. The serum and urine samples were analyzed by UHPLC-Q-TOF/MS separately.
- Group non-EA: Serum and Urine samples were collected before anesthesia and immediately after surgery from children who enrolled in part I and undergoing the adenoidectomy or adenotonsillectomy. A PAED score less than 12 was defined as non-EA. The serum and urine samples were analyzed by UHPLC-Q-TOF/MS separately.

SUMMARY:
It is known that some factors are associated with emergence agitation(EA), and investigators are still unable to predict accurately those who undergoing maxillofacial surgery are at great risks.This study intend to identify the risk factors for EA and to explore the mechanism of EA , which is helpful for early prediction, prevention and treatment in children.

DETAILED DESCRIPTION:
This study was divided into two parts. The first part, multivariate regression analysis were conducted to identify the risk factors for pain and EA following maxillofacial surgery in children. The second part, metabolomics research was used to explore the relationship between metabolites and EA in children.

ELIGIBILITY:
Eligibility Criteria in Part I

Inclusion Criteria:

1. Patients undergoing palatopharyngoplasty/tonsillar and/or adenoidectomy, auricle reconstruction, and photodynamic therapy for vascular malformations on face.
2. Aged between 3 years and 12 years.
3. American Society of Anesthesiologists(ASA) class I-II.

Exclusion Criteria:

1. Patients with developmental delays.
2. Patients with mental disorders.
3. Patients with severe liver and kidney damage,or other heart and lung disease.
4. Reject to participate in the trials.

Eligibility Criteria in Part II

Inclusion Criteria:

1. Patients who underwent adenoidectomy or adenotonsillectomy in part I of this study.
2. Aged between 3 years and 7 years.
3. American Society of Anesthesiologists(ASA) class I-II.
4. Patients who underwent sevoflurane anesthesia maintainance.

Exclusion Criteria:

1. Patients with developmental delays or mental disorders.
2. Patients with neurological or psychiatric diseases.
3. Patients with severe liver and kidney damage,or other heart and lung disease.
4. Patients with metabolic diseases or family inherited diseases.
5. Patients who received drug treatment or intravenous nutritional supports.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing palatopharyngoplasty/tonsillar and/or adenoidectomy, auricle reconstruction, and photodynamic therapy for vascular malformations on face.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Risk factors for pain and emergence agitation following maxillofacial surgery in children | within 48 hours
  Children aged 3-12 years who undergoing palatopharyngoplasty/adenoidectomy or adenotonsillectomy, auricle reconstruction, and photodynamic therapy for vascular malformations were enrolled in this study. The general information of children, preoperative anxiety state, preoperative anxiety state of parents, operation type, anesthesia method, analgesic drug, postoperative pain and emergence agitation degree were collected. Multivariate regression analysis were conducted to identify the risk factors for pain and emergence agitation following maxillofacial surgery in children.
The levels of serum and urine metabolites in EA | within 24 hours
  Children who underwent adenoidectomy or adenotonsillectomy in part I of this study were included. Urine (5ml) and peripheral venous blood (1ml) samples were collected before anesthesia and immediately after completion of agitation score. EA was defined as a Pediatric anesthesia emergence delirium(PAED) score ≥12 points. Children in EA group were matched with non-EA group, and UPLC-Q TOF/MS analysis was performed to identify the metabolites between two groups during the recovery period.

CONTACTS AND LOCATIONS:
Overall Officials: Jingjie Li, M.D, Study Chair — Shanghai No.9 People's Hospital
Locations (1):
- Shanghai No.9 People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Li J, Shi Y, Zhou X, Feng W, Han L, Ma D, Jiang H, Yuan Y. Urinary Aromatic Amino Acid Metabolites Associated With Postoperative Emergence Agitation in Paediatric Patients After General Anaesthesia: Urine Metabolomics Study. Front Pharmacol. 2022 Jul 19;13:932776. doi: 10.3389/fphar.2022.932776. eCollection 2022. PMID 35928271